CLINICAL TRIAL: NCT01315574
Title: In Vivo Effects of Antiglaucomatous Prostaglandin Therapy on Immune Cells, Epithelium, and Nerves of the Ocular Surface: A Laser In Vivo Confocal Microscopy Study
Brief Title: Effects of Anti-Glaucoma Medications on the Ocular Surface
Acronym: BAK
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow Enrollment
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-007H
Record Dates: First submitted 2011-03-10; First posted 2011-03-15 (Estimated); Results first posted 2017-02-03 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2015-01

CONDITIONS: Glaucoma
Keywords: Glaucoma; Xalatan; Travatan Z; Latanoprost; Travoprost; Dry Eye
MeSH Terms: conditions — Glaucoma; Dry Eye Syndromes | interventions — Travoprost; Latanoprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Latanoprost (Xalatan) (Active Comparator): 7 Patients were randomized to receive BAK-containing Xalatan for treatment of their glaucoma.
  Interventions: Drug: Latanoprost
- Travoprost (Travatan Z) (Active Comparator): 7 Patients were randomized to receive BAK-free Travatan Z for treatment of their glaucoma.
  Interventions: Drug: Travoprost

INTERVENTIONS:
Drug: Travoprost — One drop Travatan Z (0.004% ophthalmic solution) in affected eye once daily.
  Other Names: Travatan Z
  Arms: Travoprost (Travatan Z)
Drug: Latanoprost — One drop Xalatan (0.005% ophthalmic solution) in affected eye once daily.
  Other Names: Xalatan
  Arms: Latanoprost (Xalatan)

SUMMARY:
The purpose of the study is to compare the efficacy of FDA-approved Travoprost (Travatan Z) and Latanoprost (Xalatan)as anti-glaucoma treatment. Several studies indicate that glaucoma medications may be associated with decreased tear production and tear film break-up time (TBUT), and increased inflammatory cells in the conjunctiva (membrane lining of the eye lids and the covering of the eye) leading to dry eye. Normal tear film (coating of the eye) is continuous and blinking maintains the tear film continuity. If you keep your eyes open long enough without blinking, the tear film will start breaking up. Your eye will feel uncomfortable forcing you to blink. In patients with dry eyes, the tear film is unstable, and breaks up faster. Therefore the tear break up time in patients who have dry eyes is shorter.

In this study, the investigators will be comparing the two previously mentioned FDA-approved eye drops Latanoprost and Travoprost. The difference between the two medications is a preservative called benzalkonium chloride (BAK). Latanoprost contains BAK while Travoprost does not. The investigators will be comparing the efficacy of each medication in lowering IOP as well as trying to track the density of immune cells across the corneal surface by taking photos of your eye. The investigators will also be assessing whether either drop leads to symptoms of dry eye by comparing results from ocular surface exam tests such as TBUT.

DETAILED DESCRIPTION:
The purpose of the study is to compare the early effects of two anti-glaucoma eye drops on eye pressure and inflammation of the eye using a microscope. One of the eye drops contains a commonly used preservative, benzalkonium chloride (BAK), while the other is free of this preservative, instead it utilises a new ionic buffer system called SofZia. Prolonged use of BAK may be damaging to the eye surface and thus being investigated at a microscopic level in this study.

Specific aims are to assess the in vivo effect of topical BAK-containing and BAK-free prostaglandin analogue anti-glaucoma therapy on intraocular pressure (IOP), as well as on density and morphology of corneal immune cells, epithelial cells and sub-basal nerve plexus.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 years of age and may be of any race and either gender;
* Subjects must not have ever used topical prostaglandin anti-glaucomatous therapy;

  * Subject has not used anti-glaucomatous treatment in the past 30 days and has not been using prescribed anti-glaucomatous medication for more than 6 months.
  * Subject is using other topical anti-glaucomatous topical treatment and wants to switch to a prostaglandin (must have undergone 30 day washout period)
* The IRB Approved informed consent and the privacy document must be read, signed, and dated by the subject or legally authorized representative before enrollment. Additionally, the informed consent document must be signed and dated by the individual consenting the subject, as well as signed and dated by a witness, if applicable;
* Subjects must be generally healthy and have normal ocular health; and
* Subjects must be willing to follow the study procedures and visit schedule.

Exclusion Criteria:

* Subjects must not have known sensitivities to any ingredient in any of the test articles
* Subjects must not have any systemic or ocular disease or disorder (exc refractive error), complicating factors or structural abnormality that would negatively affect the conduct or outcome of the study:

  * No prior (within 30 days of enrollment) or current ocular infections (bacterial, viral or fungal), active ocular inflammation (i.e., follicular conjunctivitis, allergic conjunctivitis, iritis), glaucoma, or preauricular lymphadenopathy.
  * No clinically significant lash or lid abnormality (e.g., trichiasis, entropion or ectropion).
  * No uncontrolled systemic disease or debilitating disease (e.g. cardiovascular disease, hypertension, diabetes, or cystic fibrosis.).
  * No prior (within 7 days of enrollment) or current, unstable active illness (e.g., upper respiratory infection).
* Pregnant woman
* Subjects must not have history of ocular surgery/trauma within the last 6 months
* Subjects must not have used any topical ocular or systemic antibiotics within 30 days of enrollment continuing throughout the study
* Subjects must not have used any topical ocular or systemic corticosteroids within 30 days of enrollment continuing throughout the study
* Subjects must not have used immunomodulator medications within 30 days of enrollment continuing throughout the study
* Subjects must not have a immune cell density of >60/fame present at their baseline confocal scan
* Subjects must not have participated in any other ophthalmic drug or device clinical trial within 30 days of enrollment.
* Inability to cooperate with the confocal exam

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pedram Hamrah, MD, Principal Investigator — Mass Eye and Ear Infirmary
Locations (1):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from May 2011 to June 2013
Period: Overall Study
Arm/Group | Latanoprost (Xalatan) | Travoprost (Travatan Z)
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: * For IOP the baseline sample size for Latanoprost is 6 patients, whereas for all other outcome measures n= 7 patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Latanoprost (Xalatan) | Travoprost (Travatan Z) | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (7.9) | 68.3 (10.0) | 66.8 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 2 | 2 | 4
Region of Enrollment [Number; unit: participants] — Participant population: newly diagnosed glaucoma patients.
  participants
    United States | 7 | 7 | 14
Central Corneal Dendritic Cell Density [Mean (Standard Deviation); unit: cells/mm^2] | 126 (88) | 91 (60) | 109 (75)
Intraocular Pressure [Mean (Standard Deviation); unit: mmHg] | 21 (6) | 22 (4) | 21.5 (4.8)
Corneal Fluorescein Staining Score [Mean (Standard Deviation); unit: units on a scale] — Corneal fluorescein staining scores range from 0 to 4 points: 0=non-staining to 4 =regional whole staining of the cornea. Higher scores indicate worse eye condition.
  units on a scale | 0.6 (1.1) | 1.3 (2.0) | 0.9 (1.6)
Tear Break-Up Time (TBUT) [Mean (Standard Deviation); unit: seconds] | 7.9 (2.0) | 8.4 (3.7) | 8.1 (2.9)

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness in Lowering Intraocular Pressure
Description: Applanation tonometry will be used to measure patients' intraocular pressure
Time Frame: At the 6 month follow-up time point
Population: Two subjects in each arm/group did not complete 6-month follow up visit. Data was not collected and analysis not completed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Latanoprost (Xalatan) | Travoprost (Travatan Z)
Number analyzed (Participants) | 5 | 5
mmHg | 13.7 (2.8) | 17.2 (2.7)

2. Secondary Outcome: Corneal Fluorescein Staining Score
Description: Corneal Fluorescein Staining score was used in this study to quantify changes in dry eye symptoms. Corneal fluorescein staining scores range from 0 to 4 points: 0=non-staining to 4 =regional whole staining of the cornea. Higher scores indicate worse eye condition.
Time Frame: At the 6 month follow-up time point
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale (1-4)
Arm/Group | Latanoprost (Xalatan) | Travoprost (Travatan Z)
Number analyzed (Participants) | 5 | 5
units on a scale (1-4) | 1 (1.7) | 1.5 (2.2)

3. Secondary Outcome: Tear Film Break-Up Time
Description: Tear Film Break-Up Time (TBUT) is a clinical test used to quantify changes in dry eye symptoms. The Tear Film Break-Up time is the number of seconds between the subjects last blink and the detection of the first dry spot in the tear film.
Time Frame: At the 6 month follow-up time point
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Latanoprost (Xalatan) | Travoprost (Travatan Z)
Number analyzed (Participants) | 5 | 5
Seconds | 6.3 (1.7) | 6.7 (3.9)

ADVERSE EVENTS:
Time Frame: Over the course of the 6 month study period
Groups:
- Travoprost (Travatan Z): 7 Patients were be randomized to receive BAK-free Travatan Z for treatment of their glaucoma.
  Travoprost: One drop Travatan Z (0.004% ophthalmic solution) in affected eye once daily.
Arm/Group | Latanoprost (Xalatan) | Travoprost (Travatan Z)
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

LIMITATIONS AND CAVEATS:
Early termination due to very slow rate of recruitment, hence reduced power of the study (small sample size); some patients lost to follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No